CLINICAL TRIAL: NCT05871684
Title: A Phase II Study of BTKi+Radiotherapy±Chemotherapy Bridging Before Chimeric Antigen Receptor T-cell Immunotherapy (CAR-T) in Combination With BTKi±PD-1 Inhibitor Maintenance Therapy for Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma (r/r B-NHL)
Brief Title: A Combination Study of CAR-T Therapy in r/r B-NHL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Prof., Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T 001
Record Dates: First submitted 2023-05-09; First posted 2023-05-23 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The combination treatment group of CAR-T therapy (Experimental): Patients dicided to receive CAR-T cell therapy will be divided into groups A and B according to their tumor burden. Group A was given a bridging regimen of BTKi (160 mg b.i.d. p.o.) + radiotherapy + chemotherapy, and group B was given a bridging regimen of BTKi (160 mg b.i.d. p.o.) + radiotherapy; BTKi (160 mg b.i.d. p.o.) was given continuously from D1 to D28 after the return of CAR-T after infusion; Based on the results of the first evaluation on day 28 after CAR-T cell infusion, CR patients were divided into groups A1 and B1, and both groups were given BTKi (160 mg b.i.d. p.o.) for 3 months maintenance; PR patients were divided into groups A2 and B2, and both groups were given BTKi (160 mg b.i.d. p.o.) for 3 months maintenance and PD-1 inhibitor (200mg q3w i.v.) for 2 years maintenance;
  Interventions: Drug: BTK inhibitor; Drug: PD-1 inhibitor

INTERVENTIONS:
Drug: BTK inhibitor — Intervention were given during bridging therapy and maintanance treament of CAR-T cell therpay.
Drug: PD-1 inhibitor — Intervention were given during maintanance treament of CAR-T cell therpay.

SUMMARY:
In registry studies of CAR-T products that have been marketed globally, patients with relapsed or refractory B-cell non-Hodgkin's lymphoma (r/r B-NHL) have been enrolled to receive CAR-T infusion in combination with tyrosine kinase inhibitors (BTKi) or immune checkpoint inhibitors (PD-1 or PD-L1 antibodies), with objective remission rate (ORR) for CAR-T in combination with BTKi ranging from 83.3%-100% and complete remission rate (CRR) were 33.3-75%. The ORRs for objective remission rates for CAR-T combined with PD1/PD-L1 ranged from 50-91% and CRRs were 33.3-64%, respectively. With regard to safety, no dose-limiting toxic (DLT) occurred and the incidence of other adverse reactions was low, and studies demonstrated that BTKi or PD-1/PD-L1 antibodies could further enhance the responsiveness and durability of anti-CD19 CAR-T cell therapy. However, there are no studies exploring the efficacy and safety of clinical regimens using BTKi + radiotherapy ± chemotherapy as a bridging regimen to treat r/r B-NHL in combination with BTKi and/or PD-1 inhibitor after CAR-T cell infusion. In real-world applications of commercial CAR-T, CAR-T therapy combined with BTKi or PD-1/PD-L1 antibodies may further improve response rates and remission persistence in r/r B-NHL patients receiving CAR-T infusion back, with efficacy benefits while ensuring a manageable safety profile. Therefore, our center plans to conduct a phase II clinical study of Regent CAR-T 001(A phase II study of BTKi+radiotherapy±chemotherapy bridging before CAR-T cell therpay in combination with BTKi±PD-1 inhibitor for r/r B-NHL).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of B-cell non-Hodgkin's lymphoma; and according to the 2014 Lugano diagnostic criteria.
* Patients who have relapsed or are refractory to at least prior first-line therapy, including anthracycline-containing chemotherapy regimens and anti-CD20 monoclonal antibody therapy; patients must meet the definitions of refractory and relapsed.
* No prior CD19 CAR-T cell therapy
* Adequate organ function to receive CAR-T cell therapy
* Vascular condition adequate to perform leukapheresis
* Able to provide written informed consent (ICF) and able to understand and agree to comply with the study requirements and assessment schedule
* Patients of childbearing potential must be willing to use highly effective contraception for the duration of the study, and for 120 days after the last dose of treatment.
* ECOG 0-2

Exclusion Criteria:

* History of allogeneic hematopoietic stem cell transplantation;
* History of epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease or any autoimmune disease involving the central nervous system;
* Presence or current concurrent other malignancies within the past 2 years, with the exception of cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors (Ta (non-invasive tumors), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane));
* Serious cardiovascular disease: grade II or higher myocardial ischemia or myocardial infarction, poorly controlled arrhythmias; grade III-IV cardiac insufficiency by NYHA criteria, or cardiac ultrasound suggestive of left ventricular ejection fraction (LVEF) <50%;
* Hypersensitivity to any study drug or excipient;
* Patients with active viral hepatitis requiring treatment as determined by the investigator: chronic hepatitis B virus carriers with HBV DNA ≥ 500 IU/mL (2500 copies/mL) (HBV DNA testing only for patients who test positive for hepatitis B surface antigen or core antibody); patients who test positive for HCV RNA (HCV testing only for patients who test positive for hepatitis C virus antibody) RNA testing);
* Patients with any active autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enterocolitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism), or a known history of allogeneic organ transplantation, or long-term heavy use of hormones or use of other immunomodulatory agents, or other patients assessed by the investigator as having implications for study treatment ;
* The presence of an active infection;
* History of uncontrollable systemic disease, including diabetes, hypertension, acute lung disease, etc;
* Known human immunodeficiency virus (HIV) infection;
* Presence of an underlying medical condition or alcohol/drug abuse or dependence that is detrimental to study drug administration, or that may affect interpretation of results, or that places the patient at high risk of developing treatment complications;
* Organ damage due to an autoimmune disease (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) or the need for systemic application of immunosuppressive or other systemic disease-controlling drugs within the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
3-month complete response rate | 3-months after CAR-T infusion
  Percentage of participants with complete response at 3-months after CAR-T infusion determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | End of treatment visit (2 years after CAR-T cell infusion)
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
1-month objective response rate | 1 month after CAR-T infusion
  Percentage of participants with response at 1-month after CAR-T infusion determined on the basis of investigator assessments according to 2014 Lugano criteria.
Progression-free survival | End of treatment visit (2 years after CAR-T cell infusion)
  Progression-free survival was defined as the time from the date of leukapheresis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall survival | End of treatment visit (2 years after CAR-T cell infusion)
  Overall survival was defined as the time from the date of leukapheresis to the date of death from any cause.
Time to reponse | End of treatment visit (2 years after CAR-T cell infusion)
  Time from CAR-T cell infusion to the first assessment of CR or PR on the basis of investigator assessments according to 2014 Lugano criteria.
Duration of response | End of treatment visit (2 years after CAR-T cell infusion)
  Time from the first efficacy assessment of CR or PR to the time of first disease progression on the basis of investigator assessments according to 2014 Lugano criteria.
Peak Plasma Concentration (Cmax) | End of treatment visit (2 years after CAR-T cell infusion)
  Detection of maximum amount of CAR-T cell expansion in patients.
Area under the plasma concentration versus time curve (AUC) | 28 days after infusion
  The area under the CAR-T concentration curve in 28 days after infusion.
Time to Peak Plasma Concentration (Tmax) | End of treatment visit (2 years after CAR-T cell infusion)
  The time to reach the highest CAR-T concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No